CLINICAL TRIAL: NCT06366945
Title: Prospective, Single-arm, Phase II Clinical Study of Tirellizumab Combined With Carboplatin and Paclitaxel Polymer Micelles Neoadjuvant Therapy for cN+ Head and Neck Squamous Cell Carcinoma
Brief Title: Tirelizumab in Combination With Carboplatin and Polymeric Micellar Paclitaxel for Neoadjuvant Therapy in cN+ HNSCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-157-02
Record Dates: First submitted 2024-04-09; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Head and Neck Cancer; HNSCC; Head Cancer Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Carboplatin; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Neoadjuvant therapy will be performed for a total of 3 cycles, with 21 days as a cycle, which includes: ① Carboplatin: AUC5, weeks 1, 3, and 6, Q3W; ② Polymeric Micellar Paclitaxel: 300mg/m2, weeks 1, 3, and 6, Q3W for three cycles; ③Tirelizumab: 200 mg weeks 1, 3, and 6, Q3W for three cycles; if adjuvant immunotherapy is omitted, Tirelizumab will be administered on weeks 1, 3, 6, 9, 12, 15 after surgery .Participants with clinical N-positive resectable head and neck squamous cell carcinoma for which standard-of-care management would entail definitive surgery followed by adjuvant radiation +/- concurrent chemotherapy are eligible.
  Interventions: Drug: Carboplatin; Drug: Tislelizumab; Drug: Polymeric Micellar Paclitaxel; Procedure: Surgical Resection of Primary +/- Neck Dissection; Radiation: Post-operative radiation therapy

INTERVENTIONS:
Drug: Carboplatin — Carboplatin AUC 5 on weeks 1, 3, and 6
Drug: Tislelizumab — Tislelizumab 200 mg on weeks 3, 6, and 9;if adjuvant immunotherapy is omitted, Tislelizumab will be administered on weeks 1, 3, 6, 9, 12, 15 after surgery
Drug: Polymeric Micellar Paclitaxel — Polymeric Micellar Paclitaxel 300mg/mg/m2 on weeks 1, 3 and 6
Procedure: Surgical Resection of Primary +/- Neck Dissection — Twenty-eight days (+ 7 days) following the 3rd cycle of neoadjuvant therapy, patients will then undergo definitive surgical resection of the primary site +/- neck dissection(s).
Radiation: Post-operative radiation therapy — Post-operative radiation therapy +/- radiosensitizing agent(s) will be administered per standard-of-care based on pathologic staging of the surgical specimen. If there is an excellent response to treatment with a high degree of downstaging the addition of adjuvant radiation may be omitted if NCCN guidelines are met. If the pathologic assesment following induction systemic therapy and surgery is ypT(pCR 或 MPR) and ypN(pCR) or ypT（ pCR 或 MPR）and ypN（ MPR）without the presence of Serious Adverse Event, adjuvant radiation will not be administered. Otherwise, patients will receive adjuvant RT-based treatment with standard radiation techniques.

SUMMARY:
To explore the efficiency and safety of Tislelizumab combinated with carboplatin and polymeric micellar paclitaxel as a new neoadjuvant treatment regimen for resectable HNSCC patients with clinical positive lymph node metastasis

DETAILED DESCRIPTION:
The 5-year overall survival rate of patients with clinical N-positive head and neck squamous cell carcinoma (HNSCC) is less than 50%, and the clinical outcomes of these patients still need improvement.

Immunotherapy, such as PD-1/PD-L1 inhibitors, has shown excellent efficiency in treating malignant tumors. Anti PD-1 therapy has been approved as a first-line treatment for recurrent/metastatic HNSCC. The results of several phase II clinical trials have shown that neoadjuvant immunotherapy for locally advanced resectable HNSCC has been proven to be safe and feasible. However, immunotherapy has a lower MPR rate for locally advanced HNSCC patients with lymph node metastasis.

Paclitaxel has been used as a first-line induction therapy for locally advanced HNSCC and is an important drug in mediating immunogenic death, enhancing the efficacy of immunotherapy. Previous studies on lung cancer have confirmed that nano-paclitaxel has better induction efficacy than solvent paclitaxel and reduces the rate of distant metastasis.

In summary, the investigators designed this study to explore the efficiency and safety of Tislelizumab combinated with carboplatin and polymeric micellar paclitaxel as a new neoadjuvant treatment regimen for patients with clinical N positive resectable HNSCC, aiming to provide a new treatment option for those patients.

ELIGIBILITY:
Inclusion Criteria:

Males and females ECOG Performance Status 0 or 1. Confirmed pathologic and/or cytologic diagnosis of squamous cell carcinoma of head and neck，T2-4N1-3M0（III-IV）（AJCC 8.0） Histological diagnosis of squamous cell carcinoma of the lip, oral cavity, oropharynx, hypopharynx, larynx.

With measurable target lesions by CT or MRI. Adequate bone marrow function. Adequate renal and liver function. Pregnancy test (for patients of childbearing potential) negative at screening. Signed Written Informed Consent.

Exclusion Criteria:

Patients who pathologically confirmed non-squamous cell carcinoma Patients who has recurrence or distant metastasis Local lesions have been surgically removed Patients who have received systemic anti-cancer therapy, including hormone therapy Patients who have received treatment targeting PD-1 or PD-L1 Patients with active autoimmune disease or a history of autoimmune disease but may relapse(Patients with the following diseases are not excluded and can be further filtered) Controlled type 1 diabetes Hypothyroidism(If it can be controlled with hormone replacement therapy) Controlled celiac disease Skin diseases that do not require systemic treatment such as Vitiligo, Psoriasis and Hair loss.

Any other disease that is not expected to recur without external triggers Any active malignant tumors within 2 years before treatment, except for the specific cancers being studied in this trial and locally recurring cancers that have been cured (such as resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical in situ Cancer or breast cancer) Any disease requiring systemic treatment with corticosteroids (referring to treatment with a dose higher than 10 mg/day of prednisone or equivalent doses of similar drugs) or other immunosuppressive treatments within 14 days before treatment.

However, patients who have currently or previously used any of the following steroid regimens can be selected:

Adrenaline replacement steroids(Prednisone ≤10mg/day or equivalent dose of similar drugs) Local, ophthalmic, intra-articular, intranasal and inhaled corticosteroids which is Systemic absorbed Minimally Prophylactically short-term (≤7 days) use of corticosteroids (for example, allergy to contrast agents) or for the treatment of non-autoimmune conditions (for example, delayed hypersensitivity reactions caused by contact allergens) Uncontrolled diabetes within 14 days before treatment or laboratory abnormalities with potassium, sodium and corrected calcium levels> 1 after standard drug treatment or hypoalbuminemia grade ≥ 3 History of the following diseases: interstitial lung disease, non-infectious pneumonia or uncontrollable diseases, including pulmonary fibrosis, acute lung disease, etc.

Severe chronic or active infection (including tuberculosis infection, etc.) that required systemic antibiotics, antibacterial or antiviral treatment occurred within 14 days before the first administration of the study drug The patient is known to have been infected with HIV Untreated patients with chronic hepatitis B or HBV carriers with chronic hepatitis B virus (HBV) DNA ≥ 500 IU/mL or active hepatitis C virus carriers (HCV) should be excluded.

Patients can be selected who is Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B patients (HBV DNA <500 IU/mL) and cured hepatitis C patients.

Any surgery requiring general anesthesia has been performed within 28 days before treatment Have had allogeneic stem cell transplantation or organ transplantation

Have any of the following cardiovascular risk factors:

Cardiogenic chest pain within 28 days before treatment(moderate pain that restricts instrumental activities of daily living) Symptomatic pulmonary embolism within 28 days before treatment Acute myocardial infarction within 6 months before treatment Any history of heart failure that has reached Grade III or IV as defined by the New York Heart Association within 6 months before treatment Grade 2 ventricular arrhythmia within 6 months before the first administration of the study drug Have a history of cerebrovascular accident within 6 months before the first administration of the study drug Have a history of severe hypersensitivity to other monoclonal antibodies Patients with treatment toxicity (caused by previous anti-cancer treatments) have not returned to baseline or stabilized, unless it is an AE that is not considered a possible safety risk (such as hair loss, neuropathy, or specific laboratory abnormalities) History of allergic reactions to cisplatin or other platinum-containing compounds Peripheral nerve disease ≥ Grade 2 defined by NCI CTCAE v5.0 standard Have gotten a live vaccine within 4 weeks before treatment(Seasonal flu vaccines are usually inactivated vaccines and are allowed to be used; The vaccine used in the nasal cavity is a live vaccine and is not allowed to be used) Abuse or dependence on alcohol or drugs and Basic medical conditions (including laboratory abnormalities) that are not conducive to the administration of the study drug , affect the interpretation of drug toxicity or AEs, lead to insufficient compliance with the study execution and possible damage The patient participates in another therapeutic clinical study at the same time

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Major pathological response (MPR) rate of metastatic lymph nodes | 10days after surgery
  the proportion of cN+ patients with the percentage of residual viable tumor cells in the tumor bed of metastatic lymph nodes less than 10%

SECONDARY OUTCOMES:
Major pathological response (MPR) rate of primary tumor | 10days after surgery
  the proportion of cN+ patients with the percentage of residual viable tumor cells in the tumor bed of primary tumors less than 10%
Event-free survival (EFS) | 1 years and 3 years
  In cancer, the length of time after primary treatment for a cancer ends that the patient remains free of certain complications or events that the treatment was intended to prevent or delay.
Overall survival（OS） | 1 years and 3 years
  The time(years) from day 1 of study treatment until death from any cause.
Incidence of treatment-related adverse events | from the first day of treatment to 30 days after surgery；if adjuvant immotherapy is omitted, time frame is from the first day of treatment to 30 days after last administration
  CTCAE 5.0
EORTC QLQ-C30 | from 1 week before treatment to 30 days after surgery
  Quality of life evaluation
pathological downstaging rate | 10days after surgery
  Percentage of patients with tumor downstaging(pathological stage≦ ypT1N0M0)
Distant metastasis-free survival(DMFS) rate | 1 year and 3 year
  The DMFS rate is evaluated and calculated from the date of random assignment until the day of first distant metastases or until the date of the last follow-up visit.
logical regional-free survival(LRFS) rate | 1 year and 3 year
  The LRFS rate is evaluated and calculated from the date of random assignment until the day of first logical regional metastases or until the date of the last follow-up visit.

OTHER OUTCOMES:
Correlation between ctDNA dynamic detection and 1-year and 2-year EFS and OS rate after Neoadjuvant immunochemotherapy | Six months after consolidation treatment
  The ctDNA dynamic detection will contain NGS test including mutations(both somatic and germline), copy number variations, gene fusions along with genetic interpretation for each and every mutation identified in each test(both blood and tissue) during the whole therapeutic process

CONTACTS AND LOCATIONS:
Overall Officials: jinsong li, doctor, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No